CLINICAL TRIAL: NCT06261606
Title: Feasibility of a Multifaceted Intervention to Mitigate the Cardiovascular Adverse Effects of Air Pollution: The COATED-AIR Feasibility Trial
Brief Title: Feasibility of a Multifaceted Program to Reduce Cardiovascular Complications of Air Pollution
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Parham Sadeghipour (Other)
Responsible Party: Sponsor-Investigator, Parham Sadeghipour, Associate professor, Rajaie Cardiovascular Medical and Research Center
Organization: Rajaie Cardiovascular Medical and Research Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 4020286
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Atherosclerosis; Coronary Artery Disease; Peripheral Arterial Disease; Ischemic Stroke; Carotid Artery Diseases
Keywords: Air Pollution; Atherosclerosis; Cardiovascular Diseases; Coronary Artery Disease; Myocardial Infarction; Peripheral Arterial Disease; Ischemic Stroke; Carotid Artery Diseases; KN-95 mask
MeSH Terms: conditions — Atherosclerosis; Coronary Artery Disease; Peripheral Arterial Disease; Ischemic Stroke; Carotid Artery Diseases; Cardiovascular Diseases; Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: Participants undergo permuted block randomization with block sizes of four via a web-based system will be used for the study, in a 1:1 ratio between the hybrid strategy or control arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hybrid strategy (Experimental): A hybrid strategy inclusive of:
  1. A one-page flashcard describing the adverse cardiovascular effects of air pollution and individual-level strategies to mitigate these effects
  2. Alerting patients on polluted days (defined as air quality index (AQI) ≥ 131 [33]) by sending cell phone text messages and recommending to not go outdoors or minimize outdoor activities (especially exercising) on those days. This will also be accompanied by periodic phone calls to ascertain that the patients receive the messages and are attentive to them.
  3. Wearing KN-95 facemasks (provided by the investigators of this study) as a physical barrier against air pollution on highly polluted days (defined as AQI ≥ 131) in case the patient cannot avoid going outdoors
  4. Dietary intervention by encouraging patients to consume citrus fruits during days with AQI ≥ 131.
  Interventions: Other: Hybrid strategy
- Usual care (No Intervention): No active strategy (usual care) without any clear recommendations related to air pollution. A control card will be shared with the patients randomized to the control group

INTERVENTIONS:
Other: Hybrid strategy — A hybrid strategy inclusive of:
  1. A one-page flashcard describing the adverse cardiovascular effects of air pollution and individual-level strategies to mitigate these effects
  2. Alerting patients on polluted days (defined as air quality index (AQI) ≥ 131 [33]) by sending cell phone text messages and recommending to not go outdoors or minimize outdoor activities (especially exercising) on those days. This will also be accompanied by periodic phone calls to ascertain that the patients receive the messages and are attentive to them.
  3. Wearing KN-95 facemasks (provided by the investigators of this study) as a physical barrier against air pollution on highly polluted days (defined as AQI ≥ 131) in case the patient cannot avoid going outdoors
  4. Dietary intervention by encouraging patients to consume citrus fruits during days with AQI ≥ 131
  Arms: Hybrid strategy

SUMMARY:
The main goal of this clinical trial is to evaluate the feasibility of conducting a large-scale clinical trial testing a program containing several aspects for reducing the effects of air pollution on cardiovascular health (which is named the hybrid program hereafter) in adult patients (18 years or older) with atherosclerotic cardiovascular disease. Furthermore, we seek to answer how much patients adhere to and are satisfied with implementing the hybrid program, and what problems executing this program will bring for patients.

DETAILED DESCRIPTION:
Background:

Air pollution, as the fourth leading cause of mortality globally, is annually responsible for 6.67 million deaths worldwide and approximately half of them are attributable to cardiovascular causes. Some of the pollutants can negatively affect the cardiovascular system, as they may pass through the lungs, entering into the bloodstream, and cause inflammation and oxidative stress. Exposure to these pollutants is associated with a diverse range of fatal and/or adverse non-fatal cardiovascular events, including myocardial infarction, heart failure, atrial fibrillation, and ischemic stroke.

Besides strategies in societal-level aiming to control the air pollution, various individual-level solutions have been suggested to mitigate the health-related effects of air pollution. Text messaging via mobile phones to alert individuals about unhealthy air quality levels, and recommending to limit activity and time spent in outdoors, use face mask when going out, or use air filtration systems are among these individual-level solutions to restrict the air pollution-related health effects. Furthermore, several studies have proposed dietary interventions and demonstrated that some nutrients, especially vitamins C and E, are potentially capable to counter with the adverse effects of air pollutants on the cardiovascular system. However, the efficacy of these individual-level solutions to reduce the the incidence of clinically relevant outcomes such as myocardial infarction, stroke, and acute limb events.

The current pilot randomized controlled trial (RCT) seeks to test the feasibility and adherence of patients with atherosclerotic cardiovascular diseases (ASCVD) to a multifaceted intervention including a one-page informational flashcard, cell phone message alerting on days with poor air quality to encourage patients not to spend time outdoors, or to wearing KN-95 facemasks outdoors in those days, and encouraging patients to consume citrus fruits on highly polluted days (which is hereafter referred to as hybrid strategy).

Randomization Procedure:

Single-center (Rajaie Cardiovascular Medical and Research Center) open-label randomized controlled trial with a 1:1 allocation ratio to hybrid strategy versus control. Permuted block randomization with block sizes of four via a web-based system will be used for the study. The specifications for the generation of the randomization schedule will be prepared by the study biostatistician. For this study, the randomization schedule refers to a list that includes the subject identification number, randomization block number, randomization code, and the allocated treatment. Such data will be kept confidential and not shared with clinical coordinators, the Steering Committee, or other trial staff members.

Outcome assessment:

The outcomes will be adjudicated by the Steering Committee, blinded to the assigned intervention

Statistical Considerations:

A convenience sample size of 50 patients (25 in the intervention arm and 25 in the control arm) is considered for this feasibility trial without power calculation for hypothesis testing. Categorical variables will be summarized as counts, percentages, and corresponding 95% confidence intervals, and will be compared between intervention and control arms using the chi-squared test. Normally distributed continuous variables will be presented as mean ± standard deviation and will be compared using the independent samples T-test. Non-normally distributed continuous variables will be expressed as median and interquartile range and will be compared using the Mann-Whitney U test. Hypothesis testing, if performed, will be for the purpose of hypothesis generation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) with documented ASCVD defined as at least one of the following:

  * Coronary artery disease (CAD):

    1. Previous or recent documented type I myocardial infarction
    2. History of coronary revascularization (percutaneous coronary intervention or coronary artery bypass graft surgery)
    3. History of obstructive CAD (>50% stenosis) documented by coronary computed tomography (CT) or conventional angiography
  * Peripheral arterial disease (PAD):

    1. Previous or recent acute ischemic limb event (>7 days prior)
    2. History of previous endovascular/surgical lower or upper extremities revascularization for an atherosclerotic cause
    3. History of ulcer or lower extremities amputation due to ASCVD.
  * Carotid arterial diseases:

    1. History of previous endovascular/surgical carotid artery revascularization for atherosclerotic cause
    2. History of > 50% carotid artery stenosis based on documented imaging tests (Duplex ultrasonography, CT angiography, magnetic resonance angiography, or conventional angiography)
  * Ischemic stroke:

    1. History of recent or previous documented ischemic stroke not due to systemic hypoperfusion/hypotension being treated with low-dose aspirin
* Willing to participate and able to provide written informed consent

Exclusion Criteria:

* Being within 7 days of acute/unstable ASCVD events (acute myocardial infarction, acute limb event, and acute ischemic stroke) or receiving triple antithrombotic therapy
* Active bleeding
* History of upper gastrointestinal bleeding within the past 30 days
* History of intracranial hemorrhage within the past 30 days
* End-stage kidney disease with estimated creatinine clearance < 15 mL/min, or undergoing hemodialysis or peritoneal dialysis
* Known aspirin sensitivity without prior successful desensitization
* Known comorbidities associated with poor prognosis (e.g., metastatic cancer) in conjunction with an estimated life expectancy of less than one year according to the treating clinician
* Vascular disease known exclusively to be from causes other than atherosclerosis (spontaneous coronary or peripheral dissection (fibromuscular dysplasia, segmental arterial mediolysis) or vasculitis such as Takayasu arteritis, Buerger's disease (i.e., thromboangiitis obliterans), and Churg Strauss syndrome
* Inherited or acquired severe coagulopathies including hemophilia and decompensated liver cirrhosis
* Any other unexpected/unwarranted conditions that make the participants unsuitable for recruitment or follow-up
* Known allergy to KN-95 or other masks, or citrus fruits
* Any facial dysmorphia that makes the patient unable or unwilling to wear a face mask
* Any medical condition necessitating unblinded facemask use for outdoor activities at the discretion of the treating clinician, or based on patient preference
* Inability to receive/read text messages/phone calls by personal mobile phone
* Unwillingness to participate, such as hesitation to wear a mask, if randomized

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-28 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility of conducting the trial | within 30 days
  Recruitment rate defined as the proportion of participants randomized divided by the proportion of eligible participants

SECONDARY OUTCOMES:
Adherence to the individual components of the hybrid strategy | within 30 days
  Adherence to any individual recommendations of the educational flashcards for mitigating the cardiovascular adverse effects of air pollution, including avoidance from going outdoors on polluted days as stated by text messaging, or wearing KN-95 facemasks if going outdoors on those days, and the dietary recommendations regarding the daily consumption of citrus fruits on highly polluted days during the 30-day follow-up. This outcome will be assessed using a custom-made questionnaire in the intervention group
Patient satisfaction with the hybrid strategy | within 30 days
  This outcome will be assessed using a custom-made 6-question questionnaire in only the intervention group, through a 5-point Likert scale for every question (1 to 5 points) with higher scores indicating better satisfaction (range= 6-30).
Any potential adverse events in intervention and control groups during the 30-day follow-up | within 30 days
  severe mask-related skin reactions, mortality (cardiovascular and non-cardiovascular), hospitalization due to cardiorespiratory causes, myocardial infarction, ischemic stroke, acute limb events, major amputation, unplanned arterial revascularization, dyspepsia and peptic ulcer disease, gastrointestinal bleeding, and major and clinically-relevant nonmajor bleeding according to International Society on Thrombosis and Haemostasis (ISTH) criteria

OTHER OUTCOMES:
Change in the health-related quality of life | within 30 days
  The change in health-related quality of life from baseline until the end of the 30-day follow-up, based on the EQ-5D-5L questionnaire, and a 5-point Likert scale for every question (1 to 5 points) with higher scores indicating better status of quality of life (range= 5-25).
Change in the level of anxiety | within 30 days
  The change in anxiety level from baseline until the end of the 30-day follow-up, based on the Generalized Anxiety Disorder-7 (GAD-7) questionnaire, and a 4-point score for every question (0 to 3 points) with higher scores indicating worse status of anxiety level (range= 5-25).

CONTACTS AND LOCATIONS:
Overall Officials: Parham Sadeghipour, M.D, Principal Investigator — Rajaie Cardiovascular Medical and Research Center
Locations (1):
- Rajaie Cardiovascular Medical and Research Center, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No